CLINICAL TRIAL: NCT00144950
Title: Urokinase Versus Primary Video-Assisted Thorascopic Surgery for Empyema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02AR04
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Empyema
MeSH Terms: conditions — Empyema

INTERVENTIONS:
Drug: insertion of a chest drain with urokinase instillation
Procedure: primary video-assisted thorascopic surgery

SUMMARY:
This study will compare VATS versus chest drain insertion and urokinase in the treatment of childhood empema by a randomised prospective study.

ELIGIBILITY:
Inclusion Criteria:

* patients under the age of 16 referred to GOSH for management of empyema

Exclusion Criteria:

-

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60

PRIMARY OUTCOMES:
length of hospital stay

SECONDARY OUTCOMES:
radiological changes at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Adam Jaffe, Dr, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Jaffe A, Calder AD, Owens CM, Stanojevic S, Sonnappa S. Role of routine computed tomography in paediatric pleural empyema. Thorax. 2008 Oct;63(10):897-902. doi: 10.1136/thx.2007.094250. Epub 2008 May 20. PMID 18492739